CLINICAL TRIAL: NCT03307655
Title: Relationship Between Nitric Oxide (NO) in Follicular Fluid and Sperm Fertilization Ability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IVI Murcia (Other)
Collaborators: Universidad de Murcia (Other); Harvard School of Public Health (HSPH) (Other); European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1602-MUR-014JL
Record Dates: First submitted 2017-10-06; First posted 2017-10-12 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Male Infertility
Keywords: nitric oxide; follicular fluid; sperm; capacitation; fertilization; phosphorylation; nitrosylation
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Intervention Model Description: Semen and FF samples will be obtained from donors and patients by masturbation after 2-7 days of sexual abstinence and they will be analyzed according to WHO guidelines (2010). FF samples will be obtained during the oocyte pick up procedure. After oocyte removal, the FF will be centrifuged for 10 min at 2000g and stored at -20°C until evaluation. NO concentration will be determined in the FF samples with the help of ion selective electrodes.
  Sperm will be capacitated in the presence and absence of FF. In a first set of experiments, the FF will be supplemented with L-Arginine and the NOS inhibitor L-NAME. In another set of experiments the same supplementations to the capacitation medium will be examined, but without using FF.
  Changes in NOS expression, protein nitrosylation, PKA activity, tyrosine phosphorylation and tyrosine nitration in sperm will be determined. The same treatment will be performed on all semen samples regardless of whether they come from patients or donors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (fertile semen donors) (Experimental): Sperm from fertile men (donors who attend the IVI Murcia clinic) will be included in this arm.
  Interventions: Other: Control (fertile semen donors)
- Patients (subfertile men) (Experimental): Sperm from patients (subfertile men, i.e. men who possess one altered spermiogram parameter, according to the WHO 2010 guidelines) will be included in this arm.
  Interventions: Other: Patients (subfertile men)

INTERVENTIONS:
Other: Control (fertile semen donors) — The sperm will be capacitated in the presence and absence of follicular fluid (FF). In a first set of experiments, the FF will be supplemented with L-Arginine and the NOS inhibitor L-NAME. In another set of experiments the same supplementations to the capacitation medium will be examined, but without using FF.
  Changes in NOS expression, protein nitrosylation, PKA activity, tyrosine phosphorylation and tyrosine nitration in sperm will be determined.
  Arms: Control (fertile semen donors)
Other: Patients (subfertile men) — The sperm will be capacitated in the presence and absence of follicular fluid (FF). In a first set of experiments, the FF will be supplemented with L-Arginine and the NOS inhibitor L-NAME. In another set of experiments the same supplementations to the capacitation medium will be examined, but without using FF.
  Changes in NOS expression, protein nitrosylation, PKA activity, tyrosine phosphorylation and tyrosine nitration in sperm will be determined.
  Arms: Patients (subfertile men)

SUMMARY:
Several studies indicate that Nitric Oxide (NO) plays an important role in the physiology of the reproductive system in mammals. It has been shown that NO affects sperm motility, it regulates the tyrosine phosphorylation of different sperm proteins, it enhances the sperm binding ability to the zona pellucida and it modulates the acrosome reaction.

The enzyme responsible for NO synthesis, the Nitric Oxide Synthase (NOS), has also been identified in the oocytes, cumulus and corona cells, as well as in the oviduct. For these reasons, the NOS presence at the fertilization site could be a key element to determine the success of this process. Therefore, carrying out in vitro studies to better understand NO's role in the fertilization process, especially in human sperm capacitation, could improve the outcome of the Assisted Reproductive Techniques (ARTs) due to an improvement both in the diagnosis of infertility and in the prognosis of treatment success.

This study is carried out in collaboration with the Animal Physiology Department from the Veterinary Faculty (University of Murcia, Spain) and it is funded by the European Commission under the Horizon 2020 Programme.

DETAILED DESCRIPTION:
Main Objective:

Determine changes in the NOS expression and protein nitrosylation in fertile and infertile patients, when adding L-Arginine, the substrate for NO synthesis, to the sperm capacitation medium in the presence/absence of human follicular fluid (hFF).

Secondary Objectives:

1. Investigate if the effects of hFF on sperm capacitation are associated to NO levels in the fluid.
2. Identify the correlation between NO levels in hFF and the clinical outcomes from ARTs.

   METHODOLOGY

   A. Population The population included in the study will comprise both semen donors and couples attending the clinic IVI Murcia for a treatment of assisted reproduction via techniques of in vitro fertilization.

   B. Inclusion / exclusion criteria Depending on the objectives, both the population and inclusion and exclusion criteria may vary.

   Inclusion criteria Main Objective

   To examine the modifications in the NOS expression as well as the protein nitrosylation in fertile and subfertile patients. For this purpose, the following groups will be recruited:
   * a group of fertile males, such as the semen donors attending the clinic IVI Murcia;
   * a group of subfertile males composed of patients, who attend the clinic IVI Murcia to undergo an in vitro fertilization treatment and who possess one altered spermiogram parameter, according to the WHO (2010) guidelines.

   In order to reach the Secondary Objectives, couples who undergo an IVF or ICSI treatment will be included.

   Exclusion criteria Will be excluded couples who undergo preimplantation genetic diagnosis, were diagnosed with repetitive abortion (three or more consecutive abortions before week 20) or implantation failure (lack of pregnancy after three embryo transfers with good quality embryos in women under 36 years of age or after two embryo transfers in women over 36 years of age), as well as women over 40 years of age.

   C. Sample size:

   Since reference values for NOS expression are not available and since the variability of the distribution of progressive spermatozoa is high, it has been determined that to detect a difference of 20% with respect to the mean in a bilateral test, with a level of significance of 5% and 80% of statistical power, 41 semen samples per group will be necessary. A period of 24 months is estimated to reach the number of seminal samples.

   D. Experimental design and interventions Biomedical research study with control group (fertile semen donors) and experimental group (subfertile males)

   Interventions:

   Semen samples: will be obtained by masturbation after 2-7 days of sexual abstinence. All samples will be analyzed according to WHO guidelines (2010). To avoid unnecessary visits for the men included in the study, the semen sample will be requested during one of their visits to the clinic.

   Spermatozoa will be capacitated in the presence and absence of hFF. In a first set of experiments, the hFF will be supplemented with L-Arginine and the NOS inhibitor L-NAME. In another set of experiments the same supplementations to the capacitation medium will be examined, but without using hFF.

   A series of techniques such as Western blot, in situ nitrosylation and Biotin Switch Assay will be used to determine any changes in the NOS expression and protein nitrosylation in spermatozoa. The Western blot technique will also be applied to evaluate other capacitation markers such as the Protein Kinase A (PKA) activity, tyrosine phosphorylation and tyrosine nitration. The same treatment will be performed on all semen samples regardless of whether they come from patients or from semen donors. IN NO CASE WILL THESE SEMEN SAMPLES BE USED TO PERFORM AN ASSISTED REPRODUCTION TREATMENT.

   Human follicular fluid samples:

   To study the correlation between the NO concentration in follicular fluid and the success of the assisted reproduction treatment, the follicular fluid samples will be obtained during the oocyte pick up procedure. After oocyte removal, these fluids are normally eliminated, but in this case the fluids will be centrifuged for 10 minutes at 2000g and stored at -20°C until evaluation.

   The NO concentration will be determined with the help of a commercially available measurement system. NO is rapidly oxidized into two stable ions, namely nitrite and nitrate, which can be assayed by using ions selective electrodes. These electrodes have been miniaturized to be able to measure samples down to 30-40 µl with detection limits down to the low µM range for both species.

   The Western blot and protein nitrosylation assays will be performed inside the Animal Physiology laboratory, at the University of Murcia (Faculty of Veterinary Medicine).

   It should be noted that the only objective of analyzing the follicular fluid is to investigate after the assisted reproduction treatment if there is any correlation between the result of the treatment and the NO levels. Under no circumstances will embryo transfer decisions be made based on the NO levels in the follicular fluid.

   E. Collection of biological samples Sperm and follicular fluid samples will be evaluated in the present study.
   * Purpose of sample collection The samples collected in the present study will only be used for the completion of the research project. To each biological sample a code will be assigned, which will be independent from the NHC code (number of clinical history) of the patients and will only be known by the research team. Dr. Juan Carlos Martínez Soto will be responsible for the storage and safekeeping of the biological samples.
   * Method for sample collection The biological samples will only be obtained once the patient has signed the corresponding informed consent. The seminal samples will be obtained by masturbation after 2-7 days of sexual abstinence. To avoid unnecessary displacements, the sample collection will take place during the visit of the patient to the clinic.

   The follicular fluid samples will be obtained on the day of the oocyte pick up procedure performed for the in vitro fertilization treatment that the patients will follow. This fluid, which is normally discarded, will be used only to determine NO values.

   Obtaining this follicular fluid does not pose any additional risk or discomfort to those caused by the reproduction treatment, since the surgical procedure of oocyte pick up is used to obtain the follicular fluid.
   * Method for sample identification The semen and follicular fluid samples will be identified in a way which will allow to safeguard the identity of the participants.
   * Sample conservation Both seminal and follicular fluid samples will be stored in freezers in the laboratory of Andrology (IVI Murcia) at -80°C until further processing, under the supervision of Dr Juan Carlos Martínez Soto. The samples sent to the University of Murcia will be stored by Dr. Carmen Matás Parra. Both the facilities of the University of Murcia and those of the IVI clinic have a restricted access, therefore the samples will be always guarded. Upon completion of the study (January 2019), the surplus samples will be destroyed following the usual protocols of the clinic.

   F. Database The data regarding sample analysis (follicular fluid and semen samples), will be stored in Excel tables in the facilities of IVI Murcia. The data regarding the results of the assisted reproduction treatments that have been followed by the patients included in the study will be obtained from the IVI management system (SIVIS).

   G. Study variables

   Four classes of variables will be distinguished according to their relevance within the study:

   Primary Variable: NO levels.

   Secondary Variables: NOS expression, rate of progressive sperm, pregnancy rate, biochemical pregnancy, pregnancy evolution, implantation rate, ectopic pregnancy rate.

   Control Variables: Tyrosine phosphorylation (optical density units), PKA (optical density units), protein nitrosylation (optical density units), nitrates and nitrites (micromolar units).

   Descriptive variables: maternal age, paternal age, male etiology, female etiology, BMI, smoking habit.

   H. Data analysis

   Descriptive analysis:

   Statistical summary of the data collected in the study. Categorical data will be presented in frequency tables and histograms. The continuous values will be summarized with the mean, standard deviation and confidence interval, they will be represented by graphs of quartiles or densities.

   The exploratory analysis of the data will allow to assess the quality of the data and the detection of anomalies.

   Analysis of homogeneity:

   The means and proportions of the descriptive variables (baseline and demographic) will be compared to validate the degree of comparability of the study groups. S chi-square test will be applied in the categorical variables and, assuming the data follow a normal distribution, a T-test in the continuous variables. If the data does not follow a normal distribution, a Mann-Whitney test would be applied.

   In the case of finding descriptive variables distributed in a way that there are statistical differences between the groups, they will be included in a regression model, to control their interference in the main relation to be studied.

   Comparison of NO expression:

   To validate a hypothesis of correlation of proportions in the NO expression, a Fisher test will be applied.

   To evaluate the effect of other covariables that can modify the behavior of NO expression, a logistic regression model will be defined.

   As for the comparison of protein nitrosylation, a Student's t-test will be applied assuming that the data follow a normal distribution. If the normality assumption will not be met, verified by a Kolmogorov-Smirnof test, a non-parametric U-MannWhitney test would be applied.

   In the same way, a linear regression model will be defined that allows the evaluation of the effect of other correlated variables.

   Evaluation of seminal quality:

   For the set of variables that make up the seminal quality, a t-Student test will be applied assuming that the data follow a normal distribution. If the normality assumption will not be met, verified by a Kolmogorov-Smirnof test, a non-parametric U-MannWhitney test would be applied.

   Evaluation of gestational outcomes:

   For the set of variables that define the gestation results, a Fisher test will be applied.

   Workplan:

   Development stages and distribution of the tasks of the entire research team, and the assignments planned for the technical staff. Indicate in addition place / center of realization of the project.

   The design of the study, as well as the drafting of the project have been carried out by Doctors Carmen Matás Parra and Juan Carlos Martínez Soto.

   The team of gynecologists who make up the Unit of Reproductive Medicine at the IVI Murcia clinic, Dr. Jose Landeras, María Nicolás, Laura Fernández and Martina Trabalón, will be responsible for the inclusion of patients and semen donors in the study, as well as the direct responsible for the assisted reproduction treatment performed on patients. Such treatment includes: the choice of treatment to be performed, ovarian stimulation, oocyte pick up procedure to collect oocytes and follicular fluid, as well as embryo transfer.

   The embryologists Marta Molla, David Gumbao, Julián Marcos, Beatriz Amorocho and Ana Isabel Sanchez will be responsible for the process of oocyte fertilization in the fertilization laboratory, as well as the selection of embryos to be transferred.

   Florentin-Daniel Staicu, Carmen Matás Parra and Juan Carlos Martínez Soto will carry out the analysis of both seminal and follicular fluid samples. These analyses will be carried out both in the facilities of the IVI Murcia clinic and in the laboratories of the University of Murcia.

   Dr. Jorge Chavarro will conduct the epidemiological and biostatistical studies.

ELIGIBILITY:
Inclusion Criteria:

* This study will include fertile males such as the semen donors attending the clinic IVI Murcia and a group of subfertile males composed of patients, who attend the clinic to undergo an in vitro fertilization treatment and who possess one altered spermiogram parameter (according to the WHO 2010 guidelines). These participants will be recruited to examine the modifications in the NOS expression as well as the protein nitrosylation in fertile and subfertile men.
* This study will also include couples who undergo an IVF or ICSI treatment, in order to investigate if the effects of human follicular fluid on sperm capacitation are associated to NO levels in the fluid and to identify the correlation between NO levels in the follicular fluid and the clinical outcomes from ARTs.

Exclusion Criteria:

* From this study will be excluded couples who undergo preimplantation genetic diagnosis, were diagnosed with repetitive abortion (three or more consecutive abortions before week 20) or implantation failure (lack of pregnancy after three embryo transfers with good quality embryos in women under 36 years of age or after two embryo transfers in women over 36 years of age), as well as women over 40 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will include: fertile and subfertile men (who will provide the semen samples) and women donors (who will provide the follicular fluid samples).
Enrollment: 82 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Nitric Oxide levels in follicular fluid | Nitrit Oxide levels will be measured within 30 min after the follicular fluid sample is available.
  Upon collection and after oocyte removal, the follicular fluid samples will be centrifuged to remove cellular debris. An aliquot will be further centrifuged in tubes with 10 kDa filters to remove proteins. This alliquot will then be used to determine NO concentration with the help of a commercially available measurement system. NO is rapidly oxidized into two stable ions, namely nitrite and nitrate, which can be assayed by using ions selective electrodes. A software will then be used to calculate the initial concentration of Nitric Oxide (micromolar).

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Matas Parra, Professor, Study Director — University of Murcia (Spain); Juan Carlos Martinez Soto, MD, PhD, Study Director — IVI Murcia (Spain); Jorge Chavarro, MD, PhD, Study Director — Harvard University; Florentin-Daniel Staicu, MSc, Principal Investigator — University of Murcia (Spain)
Locations (1):
- IVI Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
The IPD will not be shared at any point during this study. To preserve participant's anonymity, the biological samples (semen and follicular fluid) that will be collected will be identified with a code which will be different from the Number of Clinical History of the donors/patients.

REFERENCES:
- [Background] Okabe M. The cell biology of mammalian fertilization. Development. 2013 Nov;140(22):4471-9. doi: 10.1242/dev.090613. PMID 24194470
- [Background] Romero-Aguirregomezcorta J, Santa AP, Garcia-Vazquez FA, Coy P, Matas C. Nitric oxide synthase (NOS) inhibition during porcine in vitro maturation modifies oocyte protein S-nitrosylation and in vitro fertilization. PLoS One. 2014 Dec 26;9(12):e115044. doi: 10.1371/journal.pone.0115044. eCollection 2014. PMID 25542028
- [Background] Gutteridge JM, Halliwell B. Comments on review of Free Radicals in Biology and Medicine, second edition, by Barry Halliwell and John M. C. Gutteridge. Free Radic Biol Med. 1992;12(1):93-5. doi: 10.1016/0891-5849(92)90062-l. No abstract available. PMID 1537574
- [Background] Griffith OW, Stuehr DJ. Nitric oxide synthases: properties and catalytic mechanism. Annu Rev Physiol. 1995;57:707-36. doi: 10.1146/annurev.ph.57.030195.003423. No abstract available. PMID 7539994
- [Background] Snyder SH. Nitric oxide. No endothelial NO. Nature. 1995 Sep 21;377(6546):196-7. doi: 10.1038/377196a0. No abstract available. PMID 7545786
- [Background] Rosselli M, Dubey RK, Rosselli MA, Macas E, Fink D, Lauper U, Keller PJ, Imthurn B. Identification of nitric oxide synthase in human and bovine oviduct. Mol Hum Reprod. 1996 Aug;2(8):607-12. doi: 10.1093/molehr/2.8.607. PMID 9239673
- [Background] Lapointe J, Roy M, St-Pierre I, Kimmins S, Gauvreau D, MacLaren LA, Bilodeau JF. Hormonal and spatial regulation of nitric oxide synthases (NOS) (neuronal NOS, inducible NOS, and endothelial NOS) in the oviducts. Endocrinology. 2006 Dec;147(12):5600-10. doi: 10.1210/en.2005-1548. Epub 2006 Aug 24. PMID 16935840
- [Background] Reyes R, Vazquez ML, Delgado NM. Detection and bioimaging of nitric oxide in bovine oocytes and sperm cells. Arch Androl. 2004 Jul-Aug;50(4):303-9. doi: 10.1080/01485010490448471. PMID 15277009
- [Background] Tao Y, Fu Z, Zhang M, Xia G, Yang J, Xie H. Immunohistochemical localization of inducible and endothelial nitric oxide synthase in porcine ovaries and effects of NO on antrum formation and oocyte meiotic maturation. Mol Cell Endocrinol. 2004 Jul 30;222(1-2):93-103. doi: 10.1016/j.mce.2004.04.014. PMID 15249129
- [Background] Ekerhovd E, Brannstrom M, Alexandersson M, Norstrom A. Evidence for nitric oxide mediation of contractile activity in isolated strips of the human Fallopian tube. Hum Reprod. 1997 Feb;12(2):301-5. doi: 10.1093/humrep/12.2.301. PMID 9070716
- [Background] Bryant CE, Tomlinson A, Mitchell JA, Thiemermann C, Willoughby DA. Nitric oxide synthase in the rat fallopian tube is regulated during the oestrous cycle. J Endocrinol. 1995 Jul;146(1):149-57. doi: 10.1677/joe.0.1460149. PMID 7561611
- [Background] Herrero MB, Goin JC, Boquet M, Canteros MG, Franchi AM, Perez Martinez S, Polak JM, Viggiano JM, Gimeno MA. The nitric oxide synthase of mouse spermatozoa. FEBS Lett. 1997 Jul 7;411(1):39-42. doi: 10.1016/s0014-5793(97)00570-x. PMID 9247138
- [Background] Meiser H, Schulz R. Detection and localization of two constitutive NOS isoforms in bull spermatozoa. Anat Histol Embryol. 2003 Dec;32(6):321-5. doi: 10.1111/j.1439-0264.2003.00459.x. PMID 14651478
- [Background] Herrero MB, Perez Martinez S, Viggiano JM, Polak JM, de Gimeno MF. Localization by indirect immunofluorescence of nitric oxide synthase in mouse and human spermatozoa. Reprod Fertil Dev. 1996;8(5):931-4. doi: 10.1071/rd9960931. PMID 8876053
- [Background] O'Bryan MK, Zini A, Cheng CY, Schlegel PN. Human sperm endothelial nitric oxide synthase expression: correlation with sperm motility. Fertil Steril. 1998 Dec;70(6):1143-7. doi: 10.1016/s0015-0282(98)00382-3. PMID 9848308
- [Background] Hou ML, Huang SY, Lai YK, Lee WC. Geldanamycin augments nitric oxide production and promotes capacitation in boar spermatozoa. Anim Reprod Sci. 2008 Feb 1;104(1):56-68. doi: 10.1016/j.anireprosci.2007.01.006. Epub 2007 Jan 10. PMID 17280805
- [Background] Rosselli M, Imthurn B, Macas E, Keller PJ, Dubey RK. Endogenous nitric oxide modulates endothelin-1 induced contraction of bovine oviduct. Biochem Biophys Res Commun. 1994 May 30;201(1):143-8. doi: 10.1006/bbrc.1994.1680. PMID 7515230
- [Background] Miraglia E, Rullo ML, Bosia A, Massobrio M, Revelli A, Ghigo D. Stimulation of the nitric oxide/cyclic guanosine monophosphate signaling pathway elicits human sperm chemotaxis in vitro. Fertil Steril. 2007 May;87(5):1059-63. doi: 10.1016/j.fertnstert.2006.07.1540. Epub 2007 Feb 5. PMID 17280661
- [Background] Jablonka-Shariff A, Olson LM. The role of nitric oxide in oocyte meiotic maturation and ovulation: meiotic abnormalities of endothelial nitric oxide synthase knock-out mouse oocytes. Endocrinology. 1998 Jun;139(6):2944-54. doi: 10.1210/endo.139.6.6054. PMID 9607805
- [Background] Goud AP, Goud PT, Diamond MP, Abu-Soud HM. Nitric oxide delays oocyte aging. Biochemistry. 2005 Aug 30;44(34):11361-8. doi: 10.1021/bi050711f. PMID 16114873
- [Background] Schmidt HH, Gagne GD, Nakane M, Pollock JS, Miller MF, Murad F. Mapping of neural nitric oxide synthase in the rat suggests frequent co-localization with NADPH diaphorase but not with soluble guanylyl cyclase, and novel paraneural functions for nitrinergic signal transduction. J Histochem Cytochem. 1992 Oct;40(10):1439-56. doi: 10.1177/40.10.1382087.
- [Background] Cameron IT, Campbell S. Nitric oxide in the endometrium. Hum Reprod Update. 1998 Sep-Oct;4(5):565-9. doi: 10.1093/humupd/4.5.565. PMID 10027610
- [Background] Donnelly ET, Lewis SE, Thompson W, Chakravarthy U. Sperm nitric oxide and motility: the effects of nitric oxide synthase stimulation and inhibition. Mol Hum Reprod. 1997 Sep;3(9):755-62. doi: 10.1093/molehr/3.9.755. PMID 9358000
- [Background] Revelli A, Soldati G, Costamagna C, Pellerey O, Aldieri E, Massobrio M, Bosia A, Ghigo D. Follicular fluid proteins stimulate nitric oxide (NO) synthesis in human sperm: a possible role for NO in acrosomal reaction. J Cell Physiol. 1999 Jan;178(1):85-92. doi: 10.1002/(SICI)1097-4652(199901)178:13.0.CO;2-Y. PMID 9886494
- [Background] Revelli A, Costamagna C, Moffa F, Aldieri E, Ochetti S, Bosia A, Massobrio M, Lindblom B, Ghigo D. Signaling pathway of nitric oxide-induced acrosome reaction in human spermatozoa. Biol Reprod. 2001 Jun;64(6):1708-12. doi: 10.1095/biolreprod64.6.1708. PMID 11369599
- [Background] Herrero MB, de Lamirande E, Gagnon C. Nitric oxide regulates human sperm capacitation and protein-tyrosine phosphorylation in vitro. Biol Reprod. 1999 Sep;61(3):575-81. doi: 10.1095/biolreprod61.3.575. PMID 10456831
- [Background] Thundathil J, de Lamirande E, Gagnon C. Nitric oxide regulates the phosphorylation of the threonine-glutamine-tyrosine motif in proteins of human spermatozoa during capacitation. Biol Reprod. 2003 Apr;68(4):1291-8. doi: 10.1095/biolreprod.102.008276. Epub 2002 Oct 30. PMID 12606410
- [Background] Sengoku K, Tamate K, Yoshida T, Takaoka Y, Miyamoto T, Ishikawa M. Effects of low concentrations of nitric oxide on the zona pellucida binding ability of human spermatozoa. Fertil Steril. 1998 Mar;69(3):522-7. doi: 10.1016/s0015-0282(97)00537-2. PMID 9531890
- [Background] Murad F. The nitric oxide-cyclic GMP signal transduction system for intracellular and intercellular communication. Recent Prog Horm Res. 1994;49:239-48. doi: 10.1016/b978-0-12-571149-4.50016-7. PMID 7511827
- [Background] Wiesner B, Weiner J, Middendorff R, Hagen V, Kaupp UB, Weyand I. Cyclic nucleotide-gated channels on the flagellum control Ca2+ entry into sperm. J Cell Biol. 1998 Jul 27;142(2):473-84. doi: 10.1083/jcb.142.2.473. PMID 9679145
- [Background] Lohmann SM, Vaandrager AB, Smolenski A, Walter U, De Jonge HR. Distinct and specific functions of cGMP-dependent protein kinases. Trends Biochem Sci. 1997 Aug;22(8):307-12. doi: 10.1016/s0968-0004(97)01086-4. PMID 9270304
- [Background] Pfeifer A, Ruth P, Dostmann W, Sausbier M, Klatt P, Hofmann F. Structure and function of cGMP-dependent protein kinases. Rev Physiol Biochem Pharmacol. 1999;135:105-49. doi: 10.1007/BFb0033671. No abstract available. PMID 9932482
- [Background] Rahman MS, Kwon WS, Pang MG. Calcium influx and male fertility in the context of the sperm proteome: an update. Biomed Res Int. 2014;2014:841615. doi: 10.1155/2014/841615. Epub 2014 Apr 27. PMID 24877140
- [Background] Miraglia E, De Angelis F, Gazzano E, Hassanpour H, Bertagna A, Aldieri E, Revelli A, Ghigo D. Nitric oxide stimulates human sperm motility via activation of the cyclic GMP/protein kinase G signaling pathway. Reproduction. 2011 Jan;141(1):47-54. doi: 10.1530/REP-10-0151. Epub 2010 Oct 21. PMID 20965947
- [Background] Kurtz A, Gotz KH, Hamann M, Wagner C. Stimulation of renin secretion by nitric oxide is mediated by phosphodiesterase 3. Proc Natl Acad Sci U S A. 1998 Apr 14;95(8):4743-7. doi: 10.1073/pnas.95.8.4743. PMID 9539809
- [Background] Beavo JA. Cyclic nucleotide phosphodiesterases: functional implications of multiple isoforms. Physiol Rev. 1995 Oct;75(4):725-48. doi: 10.1152/physrev.1995.75.4.725. PMID 7480160
- [Background] Belen Herrero M, Chatterjee S, Lefievre L, de Lamirande E, Gagnon C. Nitric oxide interacts with the cAMP pathway to modulate capacitation of human spermatozoa. Free Radic Biol Med. 2000 Sep 15;29(6):522-36. doi: 10.1016/s0891-5849(00)00339-7. PMID 11025196
- [Background] McVey M, Hill J, Howlett A, Klein C. Adenylyl cyclase, a coincidence detector for nitric oxide. J Biol Chem. 1999 Jul 2;274(27):18887-92. doi: 10.1074/jbc.274.27.18887. PMID 10383385
- [Background] de Lamirande E, Gagnon C. The extracellular signal-regulated kinase (ERK) pathway is involved in human sperm function and modulated by the superoxide anion. Mol Hum Reprod. 2002 Feb;8(2):124-35. doi: 10.1093/molehr/8.2.124. PMID 11818515
- [Background] Lefievre L, Chen Y, Conner SJ, Scott JL, Publicover SJ, Ford WC, Barratt CL. Human spermatozoa contain multiple targets for protein S-nitrosylation: an alternative mechanism of the modulation of sperm function by nitric oxide? Proteomics. 2007 Sep;7(17):3066-84. doi: 10.1002/pmic.200700254. PMID 17683036
- [Background] Machado-Oliveira G, Lefievre L, Ford C, Herrero MB, Barratt C, Connolly TJ, Nash K, Morales-Garcia A, Kirkman-Brown J, Publicover S. Mobilisation of Ca2+ stores and flagellar regulation in human sperm by S-nitrosylation: a role for NO synthesised in the female reproductive tract. Development. 2008 Nov;135(22):3677-86. doi: 10.1242/dev.024521. Epub 2008 Oct 8. PMID 18842814
- [Background] Bedu-Addo K, Costello S, Harper C, Machado-Oliveira G, Lefievre L, Ford C, Barratt C, Publicover S. Mobilisation of stored calcium in the neck region of human sperm--a mechanism for regulation of flagellar activity. Int J Dev Biol. 2008;52(5-6):615-26. doi: 10.1387/ijdb.072535kb. PMID 18649275
- [Background] Kakizawa S, Yamazawa T, Iino M. Nitric oxide-induced calcium release: activation of type 1 ryanodine receptor by endogenous nitric oxide. Channels (Austin). 2013 Jan 1;7(1):1-5. doi: 10.4161/chan.22555. Epub 2012 Dec 17. PMID 23247505
- [Background] Takeshima H, Nishimura S, Matsumoto T, Ishida H, Kangawa K, Minamino N, Matsuo H, Ueda M, Hanaoka M, Hirose T, et al. Primary structure and expression from complementary DNA of skeletal muscle ryanodine receptor. Nature. 1989 Jun 8;339(6224):439-45. doi: 10.1038/339439a0. PMID 2725677
- [Background] Otsu K, Willard HF, Khanna VK, Zorzato F, Green NM, MacLennan DH. Molecular cloning of cDNA encoding the Ca2+ release channel (ryanodine receptor) of rabbit cardiac muscle sarcoplasmic reticulum. J Biol Chem. 1990 Aug 15;265(23):13472-83. PMID 2380170
- [Background] Rosselli M, Keller PJ, Dubey RK. Role of nitric oxide in the biology, physiology and pathophysiology of reproduction. Hum Reprod Update. 1998 Jan-Feb;4(1):3-24. doi: 10.1093/humupd/4.1.3. PMID 9622410
- [Background] Foster MW, Stamler JS. New insights into protein S-nitrosylation. Mitochondria as a model system. J Biol Chem. 2004 Jun 11;279(24):25891-7. doi: 10.1074/jbc.M313853200. Epub 2004 Apr 6. PMID 15069080
- [Background] Hess DT, Matsumoto A, Kim SO, Marshall HE, Stamler JS. Protein S-nitrosylation: purview and parameters. Nat Rev Mol Cell Biol. 2005 Feb;6(2):150-66. doi: 10.1038/nrm1569. PMID 15688001
- [Background] Morielli T, O'Flaherty C. Oxidative stress impairs function and increases redox protein modifications in human spermatozoa. Reproduction. 2015 Jan;149(1):113-23. doi: 10.1530/REP-14-0240. Epub 2014 Nov 10. PMID 25385721
- [Background] Herrero MB, de Lamirande E, Gagnon C. Tyrosine nitration in human spermatozoa: a physiological function of peroxynitrite, the reaction product of nitric oxide and superoxide. Mol Hum Reprod. 2001 Oct;7(10):913-21. doi: 10.1093/molehr/7.10.913. PMID 11574660
- [Background] Vignini A, Nanetti L, Buldreghini E, Moroni C, Ricciardo-Lamonica G, Mantero F, Boscaro M, Mazzanti L, Balercia G. The production of peroxynitrite by human spermatozoa may affect sperm motility through the formation of protein nitrotyrosine. Fertil Steril. 2006 Apr;85(4):947-53. doi: 10.1016/j.fertnstert.2005.09.027. Epub 2006 Mar 9. PMID 16580379